CLINICAL TRIAL: NCT03941496
Title: Phase 1b/2a Safety and Immunogenicity of the DNMT Inhibitor Azacitidine During Anti-Tuberculosis Therapy
Brief Title: Azacytidine During Anti-tuberculosis Therapy
Acronym: AZA
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was halted prematurely due to Bristol-Myers Squibb's (BMS) decision to withdraw support for this study.
Sponsor: Andrew Dinardo (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Andrew Dinardo, Principal Investigator / Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-45051
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Tuberculosis; TB; Mycobacterium tuberculosis; Mtb; anti-TB therapy; ATT; rifampin (R), isoniazid (H) pyrazinamide (Z) ethambutol (E); RHZE; rifampin (R), isoniazid (H); RH
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: This study is a Phase Ib/IIa single-institution, open-label, non-randomized clinical trial of using azacitidine in pulmonary TB patients during the continuation phase of ATT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZA Treatment (Experimental): In Phase Ib dose escalation stage, participants will receive subcutaneous (SQ) AZA once daily x 5 days. Results from Phase Ib are sent to FDA/IRB for approval before proceeding to Phase IIa. 36 subjects will receive AZA treatment in total (Phase Ib/IIa). All participants receive standard of care antibiotics against tuberculosis.
  Dose Escalation Strategy to identify the lowest dose of AZA that decreases DNA methylation and restores immune function is listed below. Proceeding to Phase IIa will proceed if stopping criteria are met at any of the steps below and FDA/IRB approval is obtained:
  1. 5 mg/m^2 subcutaneous (SQ) once daily x 5 days for 8 individuals
  2. 15 mg/m^2 subcutaneous (SQ) once daily x 5 days for 8 individuals
  3. 30 mg/m^2 subcutaneous (SQ) once daily x 5 days for 8 individuals
  4. 50 mg/m^2 SQ once daily x 5 days for 8 individuals
  5. 75 mg/m^2 once daily x 5 days for 8 individuals
  Interventions: Drug: Azacitidine Injection

INTERVENTIONS:
Drug: Azacitidine Injection — In Phase Ib dose escalation stage, 24 participants will receive AZA subcutaenously once a day for 5 days as follows:
  1. 5 mg/m^2
  2. 15 mg/m^2
  3. 30 mg/m^2
  4. 50 mg/m^2
  5. 75 mg/m^2
  Results from Phase Ib are sent to FDA/IRB for approval before proceeding to Phase IIa. 36 subjects will receive AZA treatment in total (Phase Ib/IIa). Subjects in Phase II will receive a dose that induces two of the three following:
  1. a decrease DNA methylation levels in genes previously identified to be persistently hyper-methylated despite successful anti-TB therapy
  2. an increase in TNF and IFN-γ signaling pathways
  3. an increase in ex vivo mycobacterial growth inhibition assay
  Other Names: AZA Group

SUMMARY:
Tuberculosis has been shown to make immune genes inaccessible and slows immune response The purpose of this research is to see if if azacitidine is safe and can return the ability of the body to resist tuberculosis (TB), a contagious infection that attacks the lungs. Individuals with tuberculosis are being asked to participate. Some will receive a drug to restore a host immunity while others can choose to receive standard of care. All patients will continue to receive standard of care tuberculosis therapy regardless of whether they chose to participate in the study.

This study is a Phase Ib/IIa single-institution, open-label, non-randomized clinical trial of sub-cutaneous azacitidine in pulmonary TB patients during the continuation phase of ATT.

DETAILED DESCRIPTION:
All study participants will have drug-sensitive TB and successfully complete 2 months of standard intensive phase 4-drug RHZE (rifampin, isoniazid, pyrazinamide, ethambutol). By definition, to have uncomplicated TB, participants will have become asymptomatic and smear-negative by the end of intense phase anti-Tb therapy and be ready to transition from standard 4-drug (INH, RIF, ETH, PZA) intense phase to the 2-drug continuation phase (INH and RIF). All participants will have 1 and 2-month cultures "no growth to date" at the time of AZA administration (1-month cultures will therefore be no growth at ~6 weeks and 2-month cultures will be no growth at ~2 weeks).

Eligible study participants will be allocated to the AZA in sequential blocks of 8 study participants.

The following will be performed during screening and work up. These procedures will be performed within 4 weeks prior to administration of study drug. A signed and dated IRB approved consent form will be obtained before study specific procedures are performed. Procedures part of routine care are not considered study specific. All subjects will be screened for eligibility before enrollment.

1. Informed consent
2. Full History and Exam

   1. Concomitant medications
   2. Allergies
   3. Alcohol and substance use
   4. Vital signs and physical exam
3. Review of baseline laboratory results including complete blood count (CBC) with differential, liver function, renal function and microbiology studies

   a. After consent, CBC, coagulation and Renal and liver function studies will occur within 14-days prior to study drug.

   i. CBC: WBC, Hemoglobin, Hematocrit, Platelet count ii. Coagulation studies: PT and PTT iii. Sodium, potassium, blood urea nitrogen, creatinine, glucose, AST, ALT, alkaline phosphatase, total bilirubin b. After screening labs, participants with cytopenias or inappropriate coagulation, renal or liver function (see inclusion and exclusion criteria), will not receive study drug
4. Pregnancy test (within 24 hours prior to AZA dosing)

PHASE IB: AZACITIDINE AFTER 10 WEEKS OF ATT; PRE-TREATMENT EVALUATION

1-Month pre-study drug: Recruitment, consent and completion of the Case Report Form (CRF) including baseline history and physical exam will occur between week 4-10 of Anti-TB therapy.

0-2 weeks pre-study drug: Blood draw for baseline immune correlates and to screen for eligibility criteria (CBC, CMP and coagulation) will occur 1-14 days prior to azacitidine dosing. A pregnancy test will occur within 24 hours prior to AZA dosing. (A CMP will include measurement of alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, total bilirubin, creatinine, chloride, carbon dioxide/bicarbonate, sodium, potassium and glucose. A CBC will include a differential and includes red blood cell count, white blood cell count, hemoglobin, hematocrit, platelet count, percent and absolute neutrophil count, percent and absolute lymphocyte count, percent and absolute monocyte count, and percent and absolute eosinophil count.)

CYCLE 1 DAYS 1-21 AZA dosing will occur during weeks 10-13 of ATT (+/- 1 week). Pretreatment enrollment labs will be reviewed, and a symptom screen and a focused exam will occur before each sub-cutaneous dosing of azacitidine. Administration includes inverting 2-3 times to homogenize contents, rolling the syringe in the palms for 30 seconds and then administering subcutaneously at a maximum of 4mL. (On subsequent days, injection sites will be > 1 inch from a previous site and only at intact and healthy skin). Subjects will come to the clinic each day (10 minute visit) for 5 days to receive the injection. A weekly telephone call will screen for symptoms with clinically relevant symptoms triggering a clinical visit and in-person evaluation.

POST DOSE FOLLOW UP Additional screenings for cytopenias, renal and liver function will occur weekly (between days 4-11, 10-18, 17-25, and 24-32). Two mL of plasma will be collected at the same time for pharmacokinetic analysis (between days 4-11, 10-18, 17-25, and 24-32). Follow up study visits and clinical evaluation will occur monthly for the last 4 months of anti-TB therapy as standard of care. Additional blood draws for PBMCs, and immune correlates will occur at week 16 of ATT (week 6 post commencing AZA).

PHASE II: AZACITIDINE AFTER 10 WEEKS OF ATT; PRE-TREATMENT EVALUATION

1-Month pre-study drug: Recruitment, consent and completion of the CRF including baseline history and physical exam will occur between week 4-10 of Anti-TB therapy.

0-2 weeks pre-study drug: Blood draw for baseline immune correlates and to screen for eligibility criteria (CBC, CMP and coagulation) will occur within 1-14 days prior to azacitidine dosing. A pregnancy test will occur within 24 hours prior to AZA dosing.

CYCLE 1 DAYS 1-21 AZA dosing will occur during weeks 10-13 of ATT (+/- 1 week). Pretreatment enrollment labs will be reviewed, and a symptom screen and a focused exam will occur before administering AZA. Subjects will come to the clinic each day (10 minute visit) for 5 days to receive the injection. A weekly telephone call will screen for symptoms with clinically relevant symptoms triggering a clinical visit and in-person evaluation.

POST DOSE FOLLOW UP Additional screenings for cytopenias, renal and liver function will occur weekly (between days 4-11, 10-18, 17-25 and 24-32). Follow up study visits and clinical evaluation will occur at week 12 (at the peak of AZA induced toxicity), 16, 20 and 24. Additional blood draws for PBMCs and immune correlates will occur at week 16 of ATT (week 6 post commencing AZA).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Microbiologically confirmed pulmonary Tuberculosis, including cavitary, lymph node or military pulmonary TB
3. Asymptomatic by the end of intense phase ATT (8 weeks) and remains asymptomatic until AZA dosing.
4. Acid-Fast Bacilli (AFB)-smear negative at the end of intensive phase.
5. 1-month sputum culture negative and 2-month sputum with no growth at time of study entry.
6. HIV-negative.
7. Adequate hepatic function (direct bilirubin 1.5 x upper limit of normal (ULN) or less, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) 1.5 x ULN or less) at the end of ATT intensive phase.
8. Adequate renal function (creatinine 2 mg/dl or less and glomular filtration rate (GFR) 60 or greater).
9. Written informed consent obtained
10. Women and men of childbearing potential must agree to use 2 clinically effective methods of contraception (e.g., oral, intrauterine device [IUD], diaphragm plus spermicide, injectable, transdermal or implantable contraception) during the study and at least 3 months after the last treatment.

Exclusion Criteria:

1. HIV-infection
2. Pre-existing liver disease as defined by imaging or pathology consistent with moderate or worse firbrosis or cirrhosis (Metavir scoring system F2)
3. Smear-positive at 2 months
4. 1-month or 2 month sputum culture positive at time of study entry.
5. Participants with extrapulmonary TB.
6. History or current drug-resistant tuberculosis
7. After consent and within two weeks before Investigational Product (IP), a study complete blood count (CBC) will be performed and individuals with cytopenias (Hemoglobin <12 g/dL, WBC < 3 cells/ mm3, Absolute Neutrophil Count (ANC) < 2,000 cells/mm3, or platelets < 110,000 platelets/mm3) will be excluded.
8. Any concurrent uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the patient at unacceptable risk of study treatment.
9. Pregnant or breast feeding females.
10. Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
11. History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie. sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity
12. Cancer (excluding surgically treated skin cancer) or hematologic malignancy currently active or active in the past three years.
13. Abnormal coagulation parameters (Prothrombin Time (PT) >15 seconds, Partial Thromboplastin (PTT) >40 seconds, and/or international normalized ratio (INR) >1.5)
14. Significant active cardiac disease within the previous 6 months including:

    1. New York Heart Association (NYHA) class 4 congestive heart failure (CHF)
    2. Unstable angina
    3. Myocardial infarction
15. Active viral infection with HIV or hepatitis type B or C
16. Known or suspected hypersensitivity to azacytidine or mannitol
17. Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of all IP-related adverse events | 2 years
  using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0.
Overall severity of all IP-related adverse events | 4 months
  using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0
Measurement of epigenetic-mediated immune exhaustion | baseline and Week 16
  measured by using 1) a standardized mycobacterial growth inhibition assay (MGIA) that measures ex vivo mycobacterial killing; 2) 18-parameter flow cytometry based multi-dimensional immune profiling (MDIP); and 3) epigenetic assays

CONTACTS AND LOCATIONS:
Overall Officials: Andrew DiNardo, Principal Investigator — Baylor College of Medicine
Locations (1):
- Harris Health System - Ben Taub Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiNardo AR, Mace EM, Lesteberg K, Cirillo JD, Mandalakas AM, Graviss EA, Orange JS, Makedonas G. Schistosome Soluble Egg Antigen Decreases Mycobacterium tuberculosis-Specific CD4+ T-Cell Effector Function With Concomitant Arrest of Macrophage Phago-Lysosome Maturation. J Infect Dis. 2016 Aug 1;214(3):479-88. doi: 10.1093/infdis/jiw156. Epub 2016 Apr 18. PMID 27389351
- [Background] Starke JR. Mortality in childhood tuberculosis: has there been progress? Lancet Infect Dis. 2017 Mar;17(3):239-241. doi: 10.1016/S1473-3099(16)30537-0. Epub 2016 Dec 8. No abstract available. PMID 27964821
- [Background] van der Walt M, Lancaster J, Shean K. Tuberculosis Case Fatality and Other Causes of Death among Multidrug-Resistant Tuberculosis Patients in a High HIV Prevalence Setting, 2000-2008, South Africa. PLoS One. 2016 Mar 7;11(3):e0144249. doi: 10.1371/journal.pone.0144249. eCollection 2016. PMID 26950554
- [Background] Bustamante J, Boisson-Dupuis S, Abel L, Casanova JL. Mendelian susceptibility to mycobacterial disease: genetic, immunological, and clinical features of inborn errors of IFN-gamma immunity. Semin Immunol. 2014 Dec;26(6):454-70. doi: 10.1016/j.smim.2014.09.008. Epub 2014 Oct 26. PMID 25453225
- [Background] DiNardo AR, Rajapakshe K, Nishiguchi T, Grimm SL, Mtetwa G, Dlamini Q, Kahari J, Mahapatra S, Kay A, Maphalala G, Mace EM, Makedonas G, Cirillo JD, Netea MG, van Crevel R, Coarfa C, Mandalakas AM. DNA hypermethylation during tuberculosis dampens host immune responsiveness. J Clin Invest. 2020 Jun 1;130(6):3113-3123. doi: 10.1172/JCI134622. PMID 32125282
- [Background] Youngblood B, Noto A, Porichis F, Akondy RS, Ndhlovu ZM, Austin JW, Bordi R, Procopio FA, Miura T, Allen TM, Sidney J, Sette A, Walker BD, Ahmed R, Boss JM, Sekaly RP, Kaufmann DE. Cutting edge: Prolonged exposure to HIV reinforces a poised epigenetic program for PD-1 expression in virus-specific CD8 T cells. J Immunol. 2013 Jul 15;191(2):540-4. doi: 10.4049/jimmunol.1203161. Epub 2013 Jun 14. PMID 23772031
- [Background] Durzynska J, Lesniewicz K, Poreba E. Human papillomaviruses in epigenetic regulations. Mutat Res Rev Mutat Res. 2017 Apr-Jun;772:36-50. doi: 10.1016/j.mrrev.2016.09.006. Epub 2016 Sep 19. PMID 28528689
- [Background] Li H, Chiappinelli KB, Guzzetta AA, Easwaran H, Yen RW, Vatapalli R, Topper MJ, Luo J, Connolly RM, Azad NS, Stearns V, Pardoll DM, Davidson N, Jones PA, Slamon DJ, Baylin SB, Zahnow CA, Ahuja N. Immune regulation by low doses of the DNA methyltransferase inhibitor 5-azacitidine in common human epithelial cancers. Oncotarget. 2014 Feb 15;5(3):587-98. doi: 10.18632/oncotarget.1782. PMID 24583822
- [Background] Mikovits JA, Young HA, Vertino P, Issa JP, Pitha PM, Turcoski-Corrales S, Taub DD, Petrow CL, Baylin SB, Ruscetti FW. Infection with human immunodeficiency virus type 1 upregulates DNA methyltransferase, resulting in de novo methylation of the gamma interferon (IFN-gamma) promoter and subsequent downregulation of IFN-gamma production. Mol Cell Biol. 1998 Sep;18(9):5166-77. doi: 10.1128/MCB.18.9.5166. PMID 9710601
- [Background] Wen H, Dou Y, Hogaboam CM, Kunkel SL. Epigenetic regulation of dendritic cell-derived interleukin-12 facilitates immunosuppression after a severe innate immune response. Blood. 2008 Feb 15;111(4):1797-804. doi: 10.1182/blood-2007-08-106443. Epub 2007 Nov 30. PMID 18055863
- [Background] Sahiratmadja E, Alisjahbana B, de Boer T, Adnan I, Maya A, Danusantoso H, Nelwan RH, Marzuki S, van der Meer JW, van Crevel R, van de Vosse E, Ottenhoff TH. Dynamic changes in pro- and anti-inflammatory cytokine profiles and gamma interferon receptor signaling integrity correlate with tuberculosis disease activity and response to curative treatment. Infect Immun. 2007 Feb;75(2):820-9. doi: 10.1128/IAI.00602-06. Epub 2006 Dec 4. PMID 17145950
- [Background] Zumla A, Rao M, Dodoo E, Maeurer M. Potential of immunomodulatory agents as adjunct host-directed therapies for multidrug-resistant tuberculosis. BMC Med. 2016 Jun 15;14:89. doi: 10.1186/s12916-016-0635-1. PMID 27301245
- [Background] Tough DF, Tak PP, Tarakhovsky A, Prinjha RK. Epigenetic drug discovery: breaking through the immune barrier. Nat Rev Drug Discov. 2016 Dec;15(12):835-853. doi: 10.1038/nrd.2016.185. Epub 2016 Oct 21. PMID 27765940
- [Background] Maio M, Covre A, Fratta E, Di Giacomo AM, Taverna P, Natali PG, Coral S, Sigalotti L. Molecular Pathways: At the Crossroads of Cancer Epigenetics and Immunotherapy. Clin Cancer Res. 2015 Sep 15;21(18):4040-7. doi: 10.1158/1078-0432.CCR-14-2914. PMID 26374074
- [Background] Tumes DJ, Onodera A, Suzuki A, Shinoda K, Endo Y, Iwamura C, Hosokawa H, Koseki H, Tokoyoda K, Suzuki Y, Motohashi S, Nakayama T. The polycomb protein Ezh2 regulates differentiation and plasticity of CD4(+) T helper type 1 and type 2 cells. Immunity. 2013 Nov 14;39(5):819-32. doi: 10.1016/j.immuni.2013.09.012. PMID 24238339
- [Background] Cole J, Morris P, Dickman MJ, Dockrell DH. The therapeutic potential of epigenetic manipulation during infectious diseases. Pharmacol Ther. 2016 Nov;167:85-99. doi: 10.1016/j.pharmthera.2016.07.013. Epub 2016 Aug 9. PMID 27519803
- [Background] DuPage M, Bluestone JA. Harnessing the plasticity of CD4(+) T cells to treat immune-mediated disease. Nat Rev Immunol. 2016 Mar;16(3):149-63. doi: 10.1038/nri.2015.18. Epub 2016 Feb 15. PMID 26875830
- [Background] Wrangle J, Wang W, Koch A, Easwaran H, Mohammad HP, Vendetti F, Vancriekinge W, Demeyer T, Du Z, Parsana P, Rodgers K, Yen RW, Zahnow CA, Taube JM, Brahmer JR, Tykodi SS, Easton K, Carvajal RD, Jones PA, Laird PW, Weisenberger DJ, Tsai S, Juergens RA, Topalian SL, Rudin CM, Brock MV, Pardoll D, Baylin SB. Alterations of immune response of Non-Small Cell Lung Cancer with Azacytidine. Oncotarget. 2013 Nov;4(11):2067-79. doi: 10.18632/oncotarget.1542. PMID 24162015
- [Background] Ghoneim HE, Fan Y, Moustaki A, Abdelsamed HA, Dash P, Dogra P, Carter R, Awad W, Neale G, Thomas PG, Youngblood B. De Novo Epigenetic Programs Inhibit PD-1 Blockade-Mediated T Cell Rejuvenation. Cell. 2017 Jun 29;170(1):142-157.e19. doi: 10.1016/j.cell.2017.06.007. Epub 2017 Jun 22. PMID 28648661
- [Background] Chiappinelli KB, Strissel PL, Desrichard A, Li H, Henke C, Akman B, Hein A, Rote NS, Cope LM, Snyder A, Makarov V, Budhu S, Slamon DJ, Wolchok JD, Pardoll DM, Beckmann MW, Zahnow CA, Merghoub T, Chan TA, Baylin SB, Strick R. Inhibiting DNA Methylation Causes an Interferon Response in Cancer via dsRNA Including Endogenous Retroviruses. Cell. 2015 Aug 27;162(5):974-86. doi: 10.1016/j.cell.2015.07.011. PMID 26317466
- [Background] Scarpa M, Scarpa M, Castagliuolo I, Erroi F, Basato S, Brun P, Angriman I, Castoro C. CD80 down-regulation is associated to aberrant DNA methylation in non-inflammatory colon carcinogenesis. BMC Cancer. 2016 Jul 4;16:388. doi: 10.1186/s12885-016-2405-z. PMID 27377375
- [Background] Wang LX, Mei ZY, Zhou JH, Yao YS, Li YH, Xu YH, Li JX, Gao XN, Zhou MH, Jiang MM, Gao L, Ding Y, Lu XC, Shi JL, Luo XF, Wang J, Wang LL, Qu C, Bai XF, Yu L. Low dose decitabine treatment induces CD80 expression in cancer cells and stimulates tumor specific cytotoxic T lymphocyte responses. PLoS One. 2013 May 9;8(5):e62924. doi: 10.1371/journal.pone.0062924. Print 2013. PMID 23671644
- [Background] Wang L, Amoozgar Z, Huang J, Saleh MH, Xing D, Orsulic S, Goldberg MS. Decitabine Enhances Lymphocyte Migration and Function and Synergizes with CTLA-4 Blockade in a Murine Ovarian Cancer Model. Cancer Immunol Res. 2015 Sep;3(9):1030-41. doi: 10.1158/2326-6066.CIR-15-0073. Epub 2015 Jun 8. PMID 26056145
- [Background] Laille E, Shi T, Garcia-Manero G, Cogle CR, Gore SD, Hetzer J, Kumar K, Skikne B, MacBeth KJ. Pharmacokinetics and Pharmacodynamics with Extended Dosing of CC-486 in Patients with Hematologic Malignancies. PLoS One. 2015 Aug 21;10(8):e0135520. doi: 10.1371/journal.pone.0135520. eCollection 2015. PMID 26296092
- [Background] Griffiths EA, Srivastava P, Matsuzaki J, Brumberger Z, Wang ES, Kocent J, Miller A, Roloff GW, Wong HY, Paluch BE, Lutgen-Dunckley LG, Martens BL, Odunsi K, Karpf AR, Hourigan CS, Nemeth MJ. NY-ESO-1 Vaccination in Combination with Decitabine Induces Antigen-Specific T-lymphocyte Responses in Patients with Myelodysplastic Syndrome. Clin Cancer Res. 2018 Mar 1;24(5):1019-1029. doi: 10.1158/1078-0432.CCR-17-1792. Epub 2017 Sep 25. PMID 28947565
- [Background] Vasu S, He S, Cheney C, Gopalakrishnan B, Mani R, Lozanski G, Mo X, Groh V, Whitman SP, Konopitzky R, Kossl C, Bucci D, Lucas DM, Yu J, Caligiuri MA, Blum W, Adam PJ, Borges E, Rueter B, Heider KH, Marcucci G, Muthusamy N. Decitabine enhances anti-CD33 monoclonal antibody BI 836858-mediated natural killer ADCC against AML blasts. Blood. 2016 Jun 9;127(23):2879-89. doi: 10.1182/blood-2015-11-680546. Epub 2016 Mar 24. PMID 27013443
- [Background] Chen J, Lopez-Moyado IF, Seo H, Lio CJ, Hempleman LJ, Sekiya T, Yoshimura A, Scott-Browne JP, Rao A. NR4A transcription factors limit CAR T cell function in solid tumours. Nature. 2019 Mar;567(7749):530-534. doi: 10.1038/s41586-019-0985-x. Epub 2019 Feb 27. PMID 30814732
- [Background] Martinez GJ, Pereira RM, Aijo T, Kim EY, Marangoni F, Pipkin ME, Togher S, Heissmeyer V, Zhang YC, Crotty S, Lamperti ED, Ansel KM, Mempel TR, Lahdesmaki H, Hogan PG, Rao A. The transcription factor NFAT promotes exhaustion of activated CD8(+) T cells. Immunity. 2015 Feb 17;42(2):265-278. doi: 10.1016/j.immuni.2015.01.006. Epub 2015 Feb 10. PMID 25680272
- [Background] Ahn E, Youngblood B, Lee J, Lee J, Sarkar S, Ahmed R. Demethylation of the PD-1 Promoter Is Imprinted during the Effector Phase of CD8 T Cell Exhaustion. J Virol. 2016 Sep 12;90(19):8934-46. doi: 10.1128/JVI.00798-16. Print 2016 Oct 1. PMID 27466420
- [Background] Alfei F, Kanev K, Hofmann M, Wu M, Ghoneim HE, Roelli P, Utzschneider DT, von Hoesslin M, Cullen JG, Fan Y, Eisenberg V, Wohlleber D, Steiger K, Merkler D, Delorenzi M, Knolle PA, Cohen CJ, Thimme R, Youngblood B, Zehn D. TOX reinforces the phenotype and longevity of exhausted T cells in chronic viral infection. Nature. 2019 Jul;571(7764):265-269. doi: 10.1038/s41586-019-1326-9. Epub 2019 Jun 17. PMID 31207605
- [Background] Nakayama-Hosoya K, Ishida T, Youngblood B, Nakamura H, Hosoya N, Koga M, Koibuchi T, Iwamoto A, Kawana-Tachikawa A. Epigenetic repression of interleukin 2 expression in senescent CD4+ T cells during chronic HIV type 1 infection. J Infect Dis. 2015 Jan 1;211(1):28-39. doi: 10.1093/infdis/jiu376. Epub 2014 Jul 7. PMID 25001463
- [Background] Scharer CD, Barwick BG, Youngblood BA, Ahmed R, Boss JM. Global DNA methylation remodeling accompanies CD8 T cell effector function. J Immunol. 2013 Sep 15;191(6):3419-29. doi: 10.4049/jimmunol.1301395. Epub 2013 Aug 16. PMID 23956425
- [Background] Youngblood B, Reich NO. The early expressed HIV-1 genes regulate DNMT1 expression. Epigenetics. 2008 May-Jun;3(3):149-56. doi: 10.4161/epi.3.3.6372. Epub 2008 May 31. PMID 18567946
- [Background] Botha T, Ryffel B. Reactivation of latent tuberculosis infection in TNF-deficient mice. J Immunol. 2003 Sep 15;171(6):3110-8. doi: 10.4049/jimmunol.171.6.3110. PMID 12960337
- [Background] Ehlers S. Role of tumour necrosis factor (TNF) in host defence against tuberculosis: implications for immunotherapies targeting TNF. Ann Rheum Dis. 2003 Nov;62 Suppl 2(Suppl 2):ii37-42. doi: 10.1136/ard.62.suppl_2.ii37. PMID 14532147
- [Background] Linnekamp JF, Butter R, Spijker R, Medema JP, van Laarhoven HWM. Clinical and biological effects of demethylating agents on solid tumours - A systematic review. Cancer Treat Rev. 2017 Mar;54:10-23. doi: 10.1016/j.ctrv.2017.01.004. Epub 2017 Jan 18. PMID 28189913
- [Background] Garcia-Manero G, Gore SD, Cogle C, Ward R, Shi T, Macbeth KJ, Laille E, Giordano H, Sakoian S, Jabbour E, Kantarjian H, Skikne B. Phase I study of oral azacitidine in myelodysplastic syndromes, chronic myelomonocytic leukemia, and acute myeloid leukemia. J Clin Oncol. 2011 Jun 20;29(18):2521-7. doi: 10.1200/JCO.2010.34.4226. Epub 2011 May 16. PMID 21576646
- [Background] Bernstein I, Byun HM, Mohrbacher A, Douer D, Gorospe G 3rd, Hergesheimer J, Groshen S, O'Connell C, Yang AS. A phase I biological study of azacitidine (Vidaza) to determine the optimal dose to inhibit DNA methylation. Epigenetics. 2010 Nov-Dec;5(8):750-7. doi: 10.4161/epi.5.8.13105. Epub 2010 Nov 1. PMID 20861661
- [Background] Savona MR, Kolibaba K, Conkling P, Kingsley EC, Becerra C, Morris JC, Rifkin RM, Laille E, Kellerman A, Ukrainskyj SM, Dong Q, Skikne BS. Extended dosing with CC-486 (oral azacitidine) in patients with myeloid malignancies. Am J Hematol. 2018 Oct;93(10):1199-1206. doi: 10.1002/ajh.25216. Epub 2018 Sep 3. PMID 30016552
- [Background] Wherry EJ, Kurachi M. Molecular and cellular insights into T cell exhaustion. Nat Rev Immunol. 2015 Aug;15(8):486-99. doi: 10.1038/nri3862. PMID 26205583
- [Background] Bengsch B, Johnson AL, Kurachi M, Odorizzi PM, Pauken KE, Attanasio J, Stelekati E, McLane LM, Paley MA, Delgoffe GM, Wherry EJ. Bioenergetic Insufficiencies Due to Metabolic Alterations Regulated by the Inhibitory Receptor PD-1 Are an Early Driver of CD8(+) T Cell Exhaustion. Immunity. 2016 Aug 16;45(2):358-73. doi: 10.1016/j.immuni.2016.07.008. Epub 2016 Aug 2. PMID 27496729
- [Background] Pauken KE, Sammons MA, Odorizzi PM, Manne S, Godec J, Khan O, Drake AM, Chen Z, Sen DR, Kurachi M, Barnitz RA, Bartman C, Bengsch B, Huang AC, Schenkel JM, Vahedi G, Haining WN, Berger SL, Wherry EJ. Epigenetic stability of exhausted T cells limits durability of reinvigoration by PD-1 blockade. Science. 2016 Dec 2;354(6316):1160-1165. doi: 10.1126/science.aaf2807. Epub 2016 Oct 27. PMID 27789795
- [Background] Sen DR, Kaminski J, Barnitz RA, Kurachi M, Gerdemann U, Yates KB, Tsao HW, Godec J, LaFleur MW, Brown FD, Tonnerre P, Chung RT, Tully DC, Allen TM, Frahm N, Lauer GM, Wherry EJ, Yosef N, Haining WN. The epigenetic landscape of T cell exhaustion. Science. 2016 Dec 2;354(6316):1165-1169. doi: 10.1126/science.aae0491. Epub 2016 Oct 27. PMID 27789799
- [Background] Singal R, Ramachandran K, Gordian E, Quintero C, Zhao W, Reis IM. Phase I/II study of azacitidine, docetaxel, and prednisone in patients with metastatic castration-resistant prostate cancer previously treated with docetaxel-based therapy. Clin Genitourin Cancer. 2015 Feb;13(1):22-31. doi: 10.1016/j.clgc.2014.07.008. Epub 2014 Aug 1. PMID 25178642
- [Background] Schneider BJ, Shah MA, Klute K, Ocean A, Popa E, Altorki N, Lieberman M, Schreiner A, Yantiss R, Christos PJ, Palmer R, You D, Viale A, Kermani P, Scandura JM. Phase I Study of Epigenetic Priming with Azacitidine Prior to Standard Neoadjuvant Chemotherapy for Patients with Resectable Gastric and Esophageal Adenocarcinoma: Evidence of Tumor Hypomethylation as an Indicator of Major Histopathologic Response. Clin Cancer Res. 2017 Jun 1;23(11):2673-2680. doi: 10.1158/1078-0432.CCR-16-1896. Epub 2016 Nov 10. PMID 27836862
- [Background] Juergens RA, Wrangle J, Vendetti FP, Murphy SC, Zhao M, Coleman B, Sebree R, Rodgers K, Hooker CM, Franco N, Lee B, Tsai S, Delgado IE, Rudek MA, Belinsky SA, Herman JG, Baylin SB, Brock MV, Rudin CM. Combination epigenetic therapy has efficacy in patients with refractory advanced non-small cell lung cancer. Cancer Discov. 2011 Dec;1(7):598-607. doi: 10.1158/2159-8290.CD-11-0214. Epub 2011 Nov 9. PMID 22586682
- [Background] Fu S, Hu W, Iyer R, Kavanagh JJ, Coleman RL, Levenback CF, Sood AK, Wolf JK, Gershenson DM, Markman M, Hennessy BT, Kurzrock R, Bast RC Jr. Phase 1b-2a study to reverse platinum resistance through use of a hypomethylating agent, azacitidine, in patients with platinum-resistant or platinum-refractory epithelial ovarian cancer. Cancer. 2011 Apr 15;117(8):1661-9. doi: 10.1002/cncr.25701. Epub 2010 Nov 8. PMID 21472713
- [Background] Cohen AL, Ray A, Van Brocklin M, Burnett DM, Bowen RC, Dyess DL, Butler TW, Dumlao T, Khong HT. A phase I trial of azacitidine and nanoparticle albumin bound paclitaxel in patients with advanced or metastatic solid tumors. Oncotarget. 2016 Dec 26;8(32):52413-52419. doi: 10.18632/oncotarget.14183. eCollection 2017 Aug 8. PMID 28881739
- [Background] DiNardo CD, Pratz K, Pullarkat V, Jonas BA, Arellano M, Becker PS, Frankfurt O, Konopleva M, Wei AH, Kantarjian HM, Xu T, Hong WJ, Chyla B, Potluri J, Pollyea DA, Letai A. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. Blood. 2019 Jan 3;133(1):7-17. doi: 10.1182/blood-2018-08-868752. Epub 2018 Oct 25. PMID 30361262
- [Background] Tyrrell FC, Budnick GE, Elliott T, Gillim-Ross L, Hildred MV, Mahlmeister P, Parrish N, Pentella M, Vanneste J, Wang YF, Starks AM. Probability of negative mycobacterium tuberculosis complex cultures based on time to detection of positive cultures: a multicenter evaluation of commercial-broth-based culture systems. J Clin Microbiol. 2012 Oct;50(10):3275-82. doi: 10.1128/JCM.01225-12. Epub 2012 Jul 25. PMID 22837326
- [Background] Nahid P, Dorman SE, Alipanah N, Barry PM, Brozek JL, Cattamanchi A, Chaisson LH, Chaisson RE, Daley CL, Grzemska M, Higashi JM, Ho CS, Hopewell PC, Keshavjee SA, Lienhardt C, Menzies R, Merrifield C, Narita M, O'Brien R, Peloquin CA, Raftery A, Saukkonen J, Schaaf HS, Sotgiu G, Starke JR, Migliori GB, Vernon A. Official American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America Clinical Practice Guidelines: Treatment of Drug-Susceptible Tuberculosis. Clin Infect Dis. 2016 Oct 1;63(7):e147-e195. doi: 10.1093/cid/ciw376. Epub 2016 Aug 10. PMID 27516382
- [Background] DiNardo AR, Nishiguchi T, Mace EM, Rajapakshe K, Mtetwa G, Kay A, Maphalala G, Secor WE, Mejia R, Orange JS, Coarfa C, Bhalla KN, Graviss EA, Mandalakas AM, Makedonas G. Schistosomiasis Induces Persistent DNA Methylation and Tuberculosis-Specific Immune Changes. J Immunol. 2018 Jul 1;201(1):124-133. doi: 10.4049/jimmunol.1800101. Epub 2018 May 11. PMID 29752313
- [Background] Carson WF, Cavassani KA, Dou Y, Kunkel SL. Epigenetic regulation of immune cell functions during post-septic immunosuppression. Epigenetics. 2011 Mar;6(3):273-83. doi: 10.4161/epi.6.3.14017. Epub 2011 Mar 1. PMID 21048427
- [Background] Aryee MJ, Jaffe AE, Corrada-Bravo H, Ladd-Acosta C, Feinberg AP, Hansen KD, Irizarry RA. Minfi: a flexible and comprehensive Bioconductor package for the analysis of Infinium DNA methylation microarrays. Bioinformatics. 2014 May 15;30(10):1363-9. doi: 10.1093/bioinformatics/btu049. Epub 2014 Jan 28. PMID 24478339
- [Background] Liberzon A, Birger C, Thorvaldsdottir H, Ghandi M, Mesirov JP, Tamayo P. The Molecular Signatures Database (MSigDB) hallmark gene set collection. Cell Syst. 2015 Dec 23;1(6):417-425. doi: 10.1016/j.cels.2015.12.004. PMID 26771021
- [Background] Onuchic V, Hartmaier RJ, Boone DN, Samuels ML, Patel RY, White WM, Garovic VD, Oesterreich S, Roth ME, Lee AV, Milosavljevic A. Epigenomic Deconvolution of Breast Tumors Reveals Metabolic Coupling between Constituent Cell Types. Cell Rep. 2016 Nov 15;17(8):2075-2086. doi: 10.1016/j.celrep.2016.10.057. PMID 27851969
- [Background] Lutsik P, Slawski M, Gasparoni G, Vedeneev N, Hein M, Walter J. MeDeCom: discovery and quantification of latent components of heterogeneous methylomes. Genome Biol. 2017 Mar 24;18(1):55. doi: 10.1186/s13059-017-1182-6. PMID 28340624
- [Background] Wallis RS, Vinhas SA, Johnson JL, Ribeiro FC, Palaci M, Peres RL, Sa RT, Dietze R, Chiunda A, Eisenach K, Ellner JJ. Whole blood bactericidal activity during treatment of pulmonary tuberculosis. J Infect Dis. 2003 Jan 15;187(2):270-8. doi: 10.1086/346053. Epub 2003 Jan 6. PMID 12552451
- [Background] Gurumurthy M, Verma R, Naftalin CM, Hee KH, Lu Q, Tan KH, Issac S, Lin W, Tan A, Seng KY, Lee LS, Paton NI. Activity of faropenem with and without rifampicin against Mycobacterium tuberculosis: evaluation in a whole-blood bactericidal activity trial. J Antimicrob Chemother. 2017 Jul 1;72(7):2012-2019. doi: 10.1093/jac/dkx081. PMID 28333342
- [Background] Wallis RS, Jakubiec W, Mitton-Fry M, Ladutko L, Campbell S, Paige D, Silvia A, Miller PF. Rapid evaluation in whole blood culture of regimens for XDR-TB containing PNU-100480 (sutezolid), TMC207, PA-824, SQ109, and pyrazinamide. PLoS One. 2012;7(1):e30479. doi: 10.1371/journal.pone.0030479. Epub 2012 Jan 18. PMID 22279595
- [Background] Fletcher HA, Tanner R, Wallis RS, Meyer J, Manjaly ZR, Harris S, Satti I, Silver RF, Hoft D, Kampmann B, Walker KB, Dockrell HM, Fruth U, Barker L, Brennan MJ, McShane H. Inhibition of mycobacterial growth in vitro following primary but not secondary vaccination with Mycobacterium bovis BCG. Clin Vaccine Immunol. 2013 Nov;20(11):1683-9. doi: 10.1128/CVI.00427-13. Epub 2013 Aug 28. PMID 23986316
- [Background] Jayashankar L, Hafner R. Adjunct Strategies for Tuberculosis Vaccines: Modulating Key Immune Cell Regulatory Mechanisms to Potentiate Vaccination. Front Immunol. 2016 Dec 16;7:577. doi: 10.3389/fimmu.2016.00577. eCollection 2016. PMID 28018344
- [Background] Joosten SA, van Meijgaarden KE, Arend SM, Prins C, Oftung F, Korsvold GE, Kik SV, Arts RJ, van Crevel R, Netea MG, Ottenhoff TH. Mycobacterial growth inhibition is associated with trained innate immunity. J Clin Invest. 2018 May 1;128(5):1837-1851. doi: 10.1172/JCI97508. Epub 2018 Apr 3. PMID 29461976
- [Background] Ayers M, Lunceford J, Nebozhyn M, Murphy E, Loboda A, Kaufman DR, Albright A, Cheng JD, Kang SP, Shankaran V, Piha-Paul SA, Yearley J, Seiwert TY, Ribas A, McClanahan TK. IFN-gamma-related mRNA profile predicts clinical response to PD-1 blockade. J Clin Invest. 2017 Aug 1;127(8):2930-2940. doi: 10.1172/JCI91190. Epub 2017 Jun 26. PMID 28650338
- [Background] Waddell SJ, Popper SJ, Rubins KH, Griffiths MJ, Brown PO, Levin M, Relman DA. Dissecting interferon-induced transcriptional programs in human peripheral blood cells. PLoS One. 2010 Mar 22;5(3):e9753. doi: 10.1371/journal.pone.0009753. PMID 20339534
- [Background] Verma D, Parasa VR, Raffetseder J, Martis M, Mehta RB, Netea M, Lerm M. Anti-mycobacterial activity correlates with altered DNA methylation pattern in immune cells from BCG-vaccinated subjects. Sci Rep. 2017 Sep 26;7(1):12305. doi: 10.1038/s41598-017-12110-2. PMID 28951586
- [Background] Tsai PC, Bell JT. Power and sample size estimation for epigenome-wide association scans to detect differential DNA methylation. Int J Epidemiol. 2015 Aug;44(4):1429-1441. doi: 10.1093/ije/dyv041. Epub 2015 May 13. PMID 25972603
- [Background] Cook PC, Owen H, Deaton AM, Borger JG, Brown SL, Clouaire T, Jones GR, Jones LH, Lundie RJ, Marley AK, Morrison VL, Phythian-Adams AT, Wachter E, Webb LM, Sutherland TE, Thomas GD, Grainger JR, Selfridge J, McKenzie AN, Allen JE, Fagerholm SC, Maizels RM, Ivens AC, Bird A, MacDonald AS. A dominant role for the methyl-CpG-binding protein Mbd2 in controlling Th2 induction by dendritic cells. Nat Commun. 2015 Apr 24;6:6920. doi: 10.1038/ncomms7920. PMID 25908537
- [Background] Imperial MZ, Nahid P, Phillips PPJ, Davies GR, Fielding K, Hanna D, Hermann D, Wallis RS, Johnson JL, Lienhardt C, Savic RM. A patient-level pooled analysis of treatment-shortening regimens for drug-susceptible pulmonary tuberculosis. Nat Med. 2018 Nov;24(11):1708-1715. doi: 10.1038/s41591-018-0224-2. Epub 2018 Nov 5. PMID 30397355